CLINICAL TRIAL: NCT04636853
Title: Cord Blood Platelet-rich Plasma (CB-PRP) in Retinitis Pigmentosa and Dry Age-related Macular Degeneration
Brief Title: CB-PRP in Retinitis Pigmentosa and Dry Age-related Macular Degeneration
Acronym: SiCord
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3417
Record Dates: First submitted 2020-11-14; First posted 2020-11-19 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2020-12

CONDITIONS: Retinitis Pigmentosa; Dry Age-related Macular Degeneration
Keywords: Cord blood platelet-rich plasma; Retinitis pigmentosa; Dry Age-related Macular degeneration; Macular Geographic Atrophy
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Affected Individual (Experimental): A subretinal injection of umbilical cord blood platelet-rich plasma (CB-PRP) will be performed only in one eye, the other eye will be considered as a control group.
  Interventions: Biological: Subretinal injection of umbilical cord blood platelet-rich plasma (CB-PRP)

INTERVENTIONS:
Biological: Subretinal injection of umbilical cord blood platelet-rich plasma (CB-PRP) — A subretinal injection of umbilical cord blood platelet-rich plasma (CB-PRP) will be performed only in one eye, the other eye will be considered as a control group.
  A complete morpho-functional ophthalmological evaluation will be performed in all patient at each control.

SUMMARY:
The study will provides the enrollment of patients with genetic retinal dystrophies with primary rod impairment and dry age-related macular degeneration (Geographic type) A subretinal injection of umbilical cord blood platelet-rich plasma (CB-PRP) will be performed only in one eye, the other eye will be considered as a control group.

A complete morpho-functional ophthalmological evaluation will be performed in all patients at each control.

DETAILED DESCRIPTION:
All patients underwent genetic evaluation and they reported different types of mutations that induce anatomic-functional impairment of the rods.

Patients affected by bilateral dry age-related macular degeneration (Geographic type) will be recruited as well.

After selecting the patients to be enrolled, the study will proceed with the vitrectomy surgery and subretinal injection of umbilical cord blood platelet-rich plasma (CB-PRP) provided by the Umbilical Cord Bank according to the procedures provided for by the current legislation on blood components for non-transfusion use.

A complete ophthalmological examination will be performed at 1, 3, 6, and 12 months. They will include:

* Anterior segment biomicroscopy
* direct and indirect ophthalmoscopy
* ETDRS visual acuity assessment
* intraocular pressure measurement
* optical coherence tomography (OCT)
* OCT Angiography (OCTA)

The following assessments will be performed at baseline and at 6 and 12 months.

* Microperimetry
* Electroretinogram (ERG)
* Visually evoked potential (VEP)
* contrast sensitivity (MARS tables)
* Goldmann perimetry

Some morpho-functional data will also be collected in the contralateral eye and used as the control group.

To ensure the best safety for the patient, the first 5 eyes will be separated by a minimum of 20 days in order to observe the post-surgical evolution.

ELIGIBILITY:
Inclusion Criteria:

* Retinal dystrophies with compromised rods (only for RP patients)
* Visual Field (Manual Goldmann) V / 4e < 30 ° (only for RP patients)
* Best corrected visual acuity > Light perception
* Known genotype
* No or minimal opacity of ocular media
* No concomitant ocular (eg glaucoma, amblyopia)
* Dry Age-related Macular Degeneration (Geographic type)

Exclusion Criteria:

* Age<18 years
* Pregnancy
* Previous inflammatory / infectious events involving the eyes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Optical coherence tomography (OCT) and optical coherence tomography angiography (OCTA) morphological changes | 3 years
  Differences in structural optical coherence tomography (OCT) and OCT Angiography (OCTA) images

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Savastano, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Alfonso Savastano, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Valentini CG, Nuzzolo ER, Bianchi M, Orlando N, Iachininoto MG, Pinci P, Teofili L. Cord Blood Platelet Lysate: In Vitro Evaluation to Support the Use in Regenerative Medicine. Mediterr J Hematol Infect Dis. 2019 Jan 1;11(1):e2019021. doi: 10.4084/MJHID.2019.021. eCollection 2019. PMID 30858959
- [Derived] Rizzo S, Savastano MC, Falsini B, Bernardinelli P, Boselli F, De Vico U, Carla MM, Giannuzzi F, Fossataro C, Gambini G, Crincoli E, Ferrara S, Ripa M, Killian R, Rizzo C, Valentini CG, Orlando N, Placidi G, Teofili L, Savastano A. Safety Results for Geographic Atrophy Associated with Age-Related Macular Degeneration Using Subretinal Cord Blood Platelet-Rich Plasma. Ophthalmol Sci. 2024 Jan 24;4(6):100476. doi: 10.1016/j.xops.2024.100476. eCollection 2024 Nov-Dec. PMID 39149709